CLINICAL TRIAL: NCT00859378
Title: A Prospective, Randomized Study Comparing Cemented and Non-cemented Semiendoprostheses in the Treatment of Proximal Femoral Fractures in the Elderly Patients
Brief Title: Cemented vs Non-cemented Semiendoprosthesis in the Treatment of Proximal Femoral Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: The Finnish Research Foundation for Orthopaedics and Traumatology (Unknown)
Responsible Party: Principal Investigator, Tero Yli-Kyyny, M.D., Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5203038
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hip Fracture; Proximal Femoral Fracture
Keywords: Hip; Hip endoprosthesis; Hip fracture; Femoral fracture; Bone cement; Non-cemented
MeSH Terms: conditions — Hip Fractures; Proximal Femoral Fractures; Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - cemented (Active Comparator): Patients are treated with a cemented semiendoprosthesis
  Interventions: Device: Cemented semiendoprosthesis
- 2 - non-cemented (Active Comparator): Patients are treated with a non-cemented semiendoprosthesis
  Interventions: Device: non-cemented

INTERVENTIONS:
Device: Cemented semiendoprosthesis — Application of a cemented semiendoprosthesis (Basis, Smith & Nephew)
  Arms: 1 - cemented
Device: non-cemented — Patients are treated with a non-cemented semiendoprosthesis (Biomet Taperloc, Biomet Inc.)
  Arms: 2 - non-cemented

SUMMARY:
The hip semiendoprosthesis is an acceptable method to treat the proximal femoral fractures. Traditionally, the cemented version of the semiendoprosthesis has been used for this indication. However, the cementing carries a risk of fat embolism during the pressurization of the cement. The fat embolism can be avoided when using the non-cemented semiendoprosthesis. In this study we want to find out whether there are any differences in the treatment results between the cemented and non-cemented semiendoprostheses when treating the proximal femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* A proximal femoral fracture

Exclusion Criteria:

* Rheumatoid arthritis
* Pathologic fracture
* Severe dementia (preventing the informed consent)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary mortality | 3 months

SECONDARY OUTCOMES:
Prosthetic complications | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Central Hospital of North Carelia, Joensuu
  - Kuopio University Hospital, Kuopio